CLINICAL TRIAL: NCT00977522
Title: A Randomized Phase 2, Double-Blind, Placebo-Controlled, Multi-Center Study Of PF-03463275 As Add-On Therapy In Outpatients With Persistent Negative Symptoms Of Schizophrenia Treated With A Stable Dose Of A Second Generation Antipsychotic
Brief Title: A Study Of PF-03463275 As Add-On Therapy In Outpatients With Persistent Negative Symptoms Of Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9131005
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia negative symptoms adjunctive
MeSH Terms: conditions — Schizophrenia | interventions — 1-methyl-1H-imidazole-4-carboxylic acid (3-chloro-4-fluoro-benzyl)-(3-methyl-3-aza-bicyclo(3.1.0) hex-6-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03463275 (Experimental)
  Interventions: Drug: PF-03463275
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03463275 — 30 mg Controlled Release tablet BID for 12 weeks
  Arms: PF-03463275
Drug: Placebo — Placebo tablet BID
  Arms: Placebo

SUMMARY:
This study is examining the efficacy of PF-03463275 compared to placebo in treating negative symptoms of schizophrenia when added to ongoing antipsychotic treatment in stable outpatients with schizophrenia.

DETAILED DESCRIPTION:
The study was terminated on August 25, 2010 because the study's scientific validity could no longer be supported. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a current diagnosis of schizophrenia of paranoid (295.30), disorganized (295.10), or undifferentiated (295.90) subtype in the residual phase.
* Subjects must be in ongoing maintenance antipsychotic monotherapy with risperidone, olanzapine, quetiapine, ziprasidone, paliperidone, or aripiprazole. Subjects must be on a stable medication treatment regimen for at least 2 months.
* Evidence of stable symptomatology at least 3 months.

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding.
* Subjects with evidence or history of a clinically significant medical condition which would increase risk or which could interfere with the interpretation of trial results.
* Subjects who have DSM IV defined psychoactive substance dependence (including alcohol and excluding nicotine and caffeine dependence) within 12 months of screening or substance abuse within 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) Negative Subscale score | 12 weeks
Vital Signs (Blood pressure, heart rate) | 15 weeks
ECG | 15 weeks
Safety laboratory assessments | 15 weeks
Adverse events | 15 weeks

SECONDARY OUTCOMES:
Change from baseline in Quality of Life Scale (QLS) | 12 weeks
Change from baseline in MATRICS Composite Cognition Battery (MCCB) composite and individual cognition domain scores | 12 weeks
Change from baseline in PANSS Total | 12 weeks
Change from baseline in PANSS Positive Subscale | 12 weeks
Change from baseline in PANSS General Subscale | 12 weeks
Change from baseline in Clinical Global Impression Severity (CGI-S) | 12 weeks
Clinical Global Impression Improvement (CGI-I) Total Score | 12 weeks
Change from baseline in Scale for Assessment of Negative Symptoms (SANS), modified | 12 weeks
Change from baseline in Abbreviated Extrapyramidal Symptom Rating Scale | 12 weeks
Change from baseline in Global Assessment of Functioning | 12 weeks
Columbia-Suicide Severity Rating Scale (C-SSRS) | 15 weeks
Pharmacokinetic assays | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (29):
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Runnemede, New Jersey
  - Pfizer Investigational Site, Toms River, New Jersey
  - Pfizer Investigational Site, Willingboro, New Jersey
  - Pfizer Investigational Site, Fresh Meadows, New York
  - Pfizer Investigational Site, Holliswood, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Edmond, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9131005&StudyName=A%20Study%20Of%20PF-03463275%20As%20Add-On%20Therapy%20In%20Outpatients%20With%20Persistent%20Negative%20Symptoms%20Of%20Schizophrenia